CLINICAL TRIAL: NCT02828280
Title: A Comparison of Controlled Ventilation With the NuMask vs. Traditional Mask Ventilation.
Brief Title: NuMask Versus Traditional Mask Ventilation During Routine Care
Status: Completed | Type: Observational
Sponsor: Derek Sakata (Other)
Responsible Party: Sponsor-Investigator, Derek Sakata, M.D., University of Utah
Organization: University of Utah (Other)
Other Study IDs: IRB_00042299
Record Dates: First submitted 2016-06-17; First posted 2016-07-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- NuMask: Pt's randomized to Numask first will be ventilated for 10 breaths with the NuMask device first, followed by 10 breaths with the traditional face mask
  Interventions: Device: NuMask; Device: Traditional mask
- Traditional mask: patients randomized to traditional mask first will receive 10 breaths by traditional mask, followed by 10 breaths with NuMask
  Interventions: Device: NuMask; Device: Traditional mask

INTERVENTIONS:
Device: NuMask — The NuMask is a relatively new mask ventilation device that has been registered with the FDA and used in the United States since 2006.
Device: Traditional mask — A traditional air inflated facemark used to ventilate patients

SUMMARY:
The direct objective of this study is to determine whether an experienced provider can more adequately and/or easily ventilate an anesthetized patient with the NuMask device as compared to traditional bag-valve-mask ventilation. These are approved masks, being used in the patients routine care. The researchers believe that mean tidal volumes obtained by experienced providers when manually ventilating anesthetized patients with the NuMask device will be larger than when using the traditional bag-valve-mask.

ELIGIBILITY:
Inclusion Criteria:

* 44 adults total
* ASA status I-III
* aged 18-64
* elective surgery at the University of Utah under general anesthesia
* Bearded, BMI >35 or edentulous

Exclusion Criteria:

* ASA IV or higher
* Oropharyngeal or facial pathology
* Risk of aspiration (defined by need for rapid sequence intubation, uncontrolled gastroesophageal reflux disease)
* Known and/or documented difficulty placing an endotracheal tube in the past
* Limited neck extension or flexion
* Personal or familial history of malignant hyperthermia
* Known or predicted severe respiratory disease or compromise
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients selected will be undergoing elective surgery at the University of Utah
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Tidal Volume comparison | 2 minutes (one minute for NuMask, one minute for traditional mask)
  Tidal volumes delivered between the two devices will be compared

SECONDARY OUTCOMES:
Ease of use | 2 minutes
  Provider will rate each device for ease of use on a 1-5 scale with 1 being easy and 5 being difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Sakata, MD, Principal Investigator — University of Utah

REFERENCES:
- [Background] Caplan RA, Posner KL, Ward RJ, Cheney FW. Adverse respiratory events in anesthesia: a closed claims analysis. Anesthesiology. 1990 May;72(5):828-33. doi: 10.1097/00000542-199005000-00010. PMID 2339799